CLINICAL TRIAL: NCT00443053
Title: An International, Multicentre, Randomised, Double-blind, Placebo-controlled, Two-parallel Group, Phase III Study to Evaluate the Efficacy and Safety of ARIXTRA (2.5mg Subcutaneously) for the Treatment of Patients With Acute Symptomatic Isolated Superficial Thrombophlebitis of the Lower Limbs to Prevent Thromboembolic Complications
Brief Title: Evaluation Of Fondaparinux (Also Called ARIXTRA) 2.5 mg Subcutaneously Once Daily For The Treatment Of Superficial Thrombophlebitis (Also Known As Superficial Vein Thrombosis)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ART108053
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Results first posted 2010-08-02 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Thrombosis, Venous
Keywords: superficial vein thrombosis; superficial thrombophlebitis; fondaparinux; deep vein thrombosis; venous thromboembolism treatment; thrombosis
MeSH Terms: conditions — Venous Thrombosis; Thrombosis | interventions — Fondaparinux

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Fondaparinux 2.5mg (Active Comparator)
  Interventions: Drug: Fondaparinux 2.5mg or placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Fondaparinux 2.5mg or placebo

INTERVENTIONS:
Drug: Fondaparinux 2.5mg or placebo — Fondaparinux 2.5mg or matching placebo subcutaneously once daily up to day 45 day

SUMMARY:
To evaluate fondaparinux 2.5mg subcutaneously once daily for 45 days in the treatment of acute (recent) superficial thrombophlebitis.

DETAILED DESCRIPTION:
Comparison of ARIXTRA™ in lower LImb Superficial Thrombophlebitis with placebo (CALISTO). An International, Multicentre, Randomised, Double-blind, Placebo-controlled, Two-parallel Group, Phase III Study to Evaluate the Efficacy and Safety of ARIXTRA (2.5 mg subcutaneously) for the Treatment of Patients with Acute Symptomatic Isolated Superficial Thrombophlebitis of the Lower Limbs to prevent Thromboembolic Complications

ELIGIBILITY:
Inclusion criteria:

* Acute symptomatic superficial thrombophlebitis of the lower limbs at least 5 cm long diagnosed by compression ultrasound.

Exclusion criteria:

* Superficial thrombophlebitis that is within 3 cm from the sapheno-femoral junction,
* deep vein thrombosis on ultrasound exam, deep vein thrombosis or pulmonary embolism within last 6 months, treatment for cancer during last 6 months,
* anticoagulant medication for more than 48 hours prior to inclusion,
* need for oral non-steroidal anti-inflammatory drugs during the study, significant bleeding event during past month,
* major surgery within last 3 months, low platelet count (below 100×109/L),
* kidney disease (Calculated creatinine clearance < 30 mL/min), woman of child-bearing potential not using reliable contraceptive method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3002 (Actual)
Dates: Start 2007-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (183):
- GSK Investigational Site, Sofia, Bulgaria
- Czechia (6):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Říčany
  - GSK Investigational Site, Tábor
- Estonia (3):
  - GSK Investigational Site, Saku
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (20):
  - GSK Investigational Site, Abbeville
  - GSK Investigational Site, Alès
  - GSK Investigational Site, Amiens
  - GSK Investigational Site, Annecy
  - GSK Investigational Site, Annonay
  - GSK Investigational Site, Arras
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Saint-Aubin-sur-Scie
  - GSK Investigational Site, Saint-Priest-en-Jarez
  - GSK Investigational Site, Tarbes
  - GSK Investigational Site, Toulon
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Valenciennes
  - GSK Investigational Site, Villeurbanne
- Germany (45):
  - GSK Investigational Site, Baesweiler, Baden-Wurttemberg
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Karlsbad, Baden-Wurttemberg
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Lauffen am Neckar, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Großheirath, Bavaria
  - GSK Investigational Site, Hemau, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Mühldorf, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Dahlwitz-Hoppegarten, Brandenburg
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Darmstadt, Hesse
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Bad Bevensen, Lower Saxony
  - GSK Investigational Site, Leer, Lower Saxony
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Kettwig, North Rhine-Westphalia
  - GSK Investigational Site, Koeln-Junkersdorf, North Rhine-Westphalia
  - GSK Investigational Site, Mönchengladbach, North Rhine-Westphalia
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Oberhausen, North Rhine-Westphalia
  - GSK Investigational Site, Waldbröl, North Rhine-Westphalia
  - GSK Investigational Site, Wuppertal, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Neustadt, Rhineland-Palatinate
  - GSK Investigational Site, Neunkirchen, Saarland
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Kirchberg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Altenburg, Thuringia
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Nordhausen, Thuringia
- Greece (6):
  - GSK Investigational Site, Alexandroupoli
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Melissia Athens
  - GSK Investigational Site, Thessaloniki
- Hungary (12):
  - GSK Investigational Site, Békéscsaba
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Esztergom
  - GSK Investigational Site, Gyula
  - GSK Investigational Site, Kaposvár
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Nyiregyháza
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Székesfehérvár
  - GSK Investigational Site, Szikszó
  - GSK Investigational Site, Zalaegerszeg
- Israel (7):
  - GSK Investigational Site, Afula
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Safed
  - GSK Investigational Site, Tel Aviv
- Italy (11):
  - GSK Investigational Site, Chieti Scalo, Abruzzo
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Piacenza, Emilia-Romagna
  - GSK Investigational Site, Reggio Emilia, Emilia-Romagna
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Padua, Veneto
  - GSK Investigational Site, Venezia, Veneto
- Latvia (2):
  - GSK Investigational Site, Daugavpils
  - GSK Investigational Site, Riga
- Netherlands (5):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Weerselo
- Poland (6):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gniewkowo
  - GSK Investigational Site, Grudziądz
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Wroclaw
- Russia (21):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Kursk
  - GSK Investigational Site, Lipetsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Rostov-on-Don
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saint Petersburgh
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Stavropol
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Tyumen
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- Slovakia (6):
  - GSK Investigational Site, Bardejov
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Nitra
  - GSK Investigational Site, Prešov
  - GSK Investigational Site, Žilina
- Spain (15):
  - GSK Investigational Site, Ávila
  - GSK Investigational Site, Boadilla Del Monte (Madrid)
  - GSK Investigational Site, Cartagena (Murcia)
  - GSK Investigational Site, Getafe
  - GSK Investigational Site, Gijón
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Mataró
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, Sant Joan d'Alacant
  - GSK Investigational Site, Segovia
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Zamora
- Switzerland (7):
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Bruderholz
  - GSK Investigational Site, Fribourg
  - GSK Investigational Site, Geneva
  - GSK Investigational Site, Lausanne
  - GSK Investigational Site, Lucerne
  - GSK Investigational Site, Zurich
- Ukraine (10):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Sevastopol
  - GSK Investigational Site, Uzhhorod
  - GSK Investigational Site, Vinnitsa
  - GSK Investigational Site, Zaporizhzhya

REFERENCES:
- [Derived] Leizorovicz A, Becker F, Buchmuller A, Quere I, Prandoni P, Decousus H; CALISTO Study Group. Clinical relevance of symptomatic superficial-vein thrombosis extension: lessons from the CALISTO study. Blood. 2013 Sep 5;122(10):1724-9. doi: 10.1182/blood-2013-04-498014. Epub 2013 Jul 2. PMID 23821661
- [Derived] Decousus H, Prandoni P, Mismetti P, Bauersachs RM, Boda Z, Brenner B, Laporte S, Matyas L, Middeldorp S, Sokurenko G, Leizorovicz A; CALISTO Study Group. Fondaparinux for the treatment of superficial-vein thrombosis in the legs. N Engl J Med. 2010 Sep 23;363(13):1222-32. doi: 10.1056/NEJMoa0912072. PMID 20860504

RESULTS

PARTICIPANT FLOW:
Groups:
- Fondaparinux 2.5 mg: Fondaparinux 2.5 milligrams (mg) administered subcutaneously (SC) once daily for 45 days
- Placebo: Matching placebo
Period: Overall Study
Arm/Group | Fondaparinux 2.5 mg | Placebo
Started | 1502 | 1500
Completed | 1481 | 1467
Not Completed | 21 | 33
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 9 | 18
Not completed — Lost to Follow-up | 4 | 5
Not completed — Did Not Meet Eligibility Criteria | 1 | 0
Not completed — Noncompliance | 2 | 1
Not completed — Other | 3 | 4
Not completed — Physician Decision | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fondaparinux 2.5 mg | Placebo | Total
Number analyzed (Participants) | 1502 | 1500 | 3002
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (13.29) | 56.9 (13.56) | 57.0 (13.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 974 | 944 | 1918
  Male | 528 | 556 | 1084
Race/Ethnicity, Customized [Number; unit: participants]
  White, European Heritage | 1485 | 1492 | 2977
  Arabic/North African Heritage | 15 | 4 | 19
  African American Heritage | 0 | 2 | 2
  Asian/South Asian Heritage | 0 | 1 | 1
  Mixed Race | 1 | 0 | 1
  Missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least on Event of Venous Thromboembolism (VTE) and/or Death From Any Cause Recorded up to Day 47
Description: VTE was defined as a composite of symptomatic deep-vein thrombosis (DVT), symptomatic pulmonary embolism (PE), symptomatic extension of superficial vein thrombosis (SVT), or symptomatic recurrence of SVT. All VTEs were confirmed by objective tests and then adjudicated by an independent central adjudication committee (CAC), whose members were blinded to treatment assignment.
Time Frame: Baseline to Day 47
Population: Intent-to-Treat (ITT) Population: all randomized participants
Measure: Number; unit: participants
Arm/Group | Fondaparinux 2.5 mg | Placebo
Number analyzed (Participants) | 1502 | 1500
participants | 13 | 88
Statistical Analysis 1: Comparison: Fondaparinux 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact; Risk Ratio (RR) = 0.15, 95% CI 2-sided [0.08 to 0.26]

2. Secondary Outcome: Number of Participants With at Least One Event of Venous Thromboembolism (VTE) and/or Death From Any Cause Recorded up to Day 77
Description: as for outcome 1
Time Frame: Baseline to Day 77
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Fondaparinux 2.5 mg | Placebo
Number analyzed (Participants) | 1502 | 1500
participants | 18 | 94
Statistical Analysis 1: Comparison: Fondaparinux 2.5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact; Risk Ratio (RR) = 0.19, 95% CI 2-sided [0.12 to 0.32]

3. Secondary Outcome: Number of Participants With at Least One Occurrence of Each Adjudicated Component of the Primary Efficacy Endpoint at Days (D) 47 and 77
Description: VTE was defined as a composite of symptomatic DVT; symptomatic PE; symptomatic extension of SVT, defined as downstream progression of the initial SVT by at least 2 cm and to within <=3 cm from the sapheno-femoral junction; or symptomatic recurrence of SVT, defined as a new episode in any other superficial venous location, meeting the following criteria: the new SVT was in a different superficial vein and not directly contiguous upstream with the index SVT, or it was in the same superficial vein but clearly distinct from the index SVT with an open venous segment of at least 10 cm in length.
Time Frame: Days 47 and 77
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Fondaparinux 2.5 mg | Placebo
Number analyzed (Participants) | 1502 | 1500
participants
  Participants with at least one event, D 47 | 13 | 88
  Death, D 47 | 2 | 1
  Symptomatic PE, D 47 | 0 | 5
  Symptomatic DVT, D 47 | 3 | 18
  Symptomatic recurrence of SVT, D 47 | 5 | 24
  Symptomatic extension of SVT, D 47 | 4 | 51
  Participants with at least one event, D 77 | 18 | 94
  Death, D 77 | 2 | 1
  Symptomatic PE, D 77 | 0 | 6
  Symptomatic DVT, D 77 | 4 | 19
  Symptomatic recurrence of SVT, D 77 | 8 | 26
  Symptomatic extension of SVT, D 77 | 5 | 54

4. Secondary Outcome: Number of Participants Who Required Surgery to Treat Superficial Vein Thrombosis Recurrence at Days 47 and 77
Description: The number of participants requiring surgery was measured.
Time Frame: Days 47 and 77
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Fondaparinux 2.5 mg | Placebo
Number analyzed (Participants) | 1502 | 1500
participants
  Day 47 | 11 | 57
  Day 77 | 15 | 61

5. Secondary Outcome: Number of Adjudicated Major Bleeding Events and Deaths at Days 47 and 77
Description: Major bleeding was defined as bleeding that was fatal and/or (1) in a critical area/organ (e.g., intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome); (2) associated with a fall in hemoglobin >=20 g/L (1.24 mmol/L); (3) led to a transfusion of >=2 units of packed red blood cells/whole blood. The revision of the Day 47 time point was to account for participants with treatment duration longer than 45 days. Adverse events were evaluated "On-Treatment," defined as from randomization up to the last injection +4 days.
Time Frame: Days 47 (or last dose plus 4 days) and 77
Population: As-Treated Population: randomized participants who received at least one dose of study treatment, as actually received
Measure: Number; unit: events
Arm/Group | Fondaparinux 2.5 mg | Placebo
Number analyzed (Participants) | 1499 | 1488
events
  Major bleeding events, Day 47 | 1 | 1
  Deaths, Day 47 | 2 | 1
  Major bleeding events, Day 77 | 1 | 1
  Deaths, Day 77 | 2 | 1

6. Secondary Outcome: Number of Adjudicated Non-Major Bleeding Events at Days 47 and 77
Description: Clinically relevant non-major bleeding was defined as clinically relevant bleeding that did not qualify as major but satisfied a priori criteria, and/or any bleeding that resulted in clinical consequences for a participant. The revision of the Day 47 time point was to account for participants with treatment duration longer than 45 days. Adverse events were evaluated "On-Treatment," defined as from randomization up to the last injection +4 days.
Time Frame: Days 47 (or last dose plus 4 days) and 77
Population: As-Treated Population
Measure: Number; unit: events
Arm/Group | Fondaparinux 2.5 mg | Placebo
Number analyzed (Participants) | 1499 | 1488
events
  Day 47 | 5 | 8
  Day 77 | 6 | 9

7. Secondary Outcome: Number of Any Adjudicated Bleeding Events at Days 47 and 77
Description: The sum of adjudicated major bleeds, non-major clinically relevant bleeds, and minor bleeds was calculated. Minor bleeding was defined as other clinically overt bleeding events that did not meet the criteria for major or clinically relevant non-major bleeding. The revision of the Day 47 time point was to account for participants with treatment duration longer than 45 days. Adverse events were evaluated "On-Treatment," defined as from randomization up to the last injection +4 days.
Time Frame: Days 47 (or last dose plus 4 days) and 77
Population: As-Treated Population
Measure: Number; unit: events
Arm/Group | Fondaparinux 2.5 mg | Placebo
Number analyzed (Participants) | 1499 | 1488
events
  Day 47 | 15 | 14
  Day 77 | 16 | 15

ADVERSE EVENTS:
Description: Serious adverse events (SAEs) and adverse events (AEs) were collected in the As-Treated Population, defined as randomized participants who received at least one dose of study treatment, as actually received.
Arm/Group | Fondaparinux 2.5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 10/1499 | 16/1488
Other Adverse Events (participants affected / at risk) | 95/1499 | 79/1488
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fondaparinux 2.5 mg (N=1499) | Placebo (N=1488)
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Billiary colic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 1
Prostatic abscess (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Vena cave thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fondaparinux 2.5 mg (N=1499) | Placebo (N=1488)
Headache (Nervous system disorders) | 34 | 31
Injection site hematoma (Skin and subcutaneous tissue disorders) | 27 | 17
Hypertension (Vascular disorders) | 20 | 15
Asthenia (General disorders) | 14 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.